CLINICAL TRIAL: NCT03471962
Title: Evaluation of Indirect Measurement of Respiratory Quotient in Non-cardiac Major Surgery as a Predictor of Anaerobic Metabolism (The BAR Study) Indirect Respiratory Quotient as a Predictor of Anaerobic Metabolism
Brief Title: Evaluation of Indirect Measurement of Respiratory Quotient in Non-cardiac Major Surgery (The BAR Study)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0006
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Surgery
Keywords: respiratory quotient (RQ); anaerobic metabolism; major surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: surgery — Indirect measurement of RQ was performed by anesthesia ventilator and compared to marker of anaerobic metabolism (arterial lactate, venoarterial PCO2 gradient, venoarterial PCO2 gradient/ arteriovenous O2 content difference, ScVO2) at different time of the srugery (every hours). In post-operative time, complications and hospital's length of stay were recorded.

SUMMARY:
Demonstrate the ability of the RQ, measured indirectly from the anesthesia ventilator, to predict the occurrence of anaerobic metabolism in patients operated of major non-cardiac surgical operation in the operating room

DETAILED DESCRIPTION:
Indirect respiratory quotient (RQ) measurement involves indirect calorimetry, which measures O2 and CO2 inspired and expired fractions. This measurement is usually used to estimate energy expenditure and which energetic substrate is preferentially used in resuscitation patients. Litterature demonstrated in a mouse model that the formation of hemorrhagic shock was associated with a change in RQ due to VCO2 and VO2 imbalance. RQ was able to distinguish anaerobic metabolism and corrected itself with correction of shock. Recently in Litterature showed a link between lactate production, cardiac output and the evolution of the RQ measured by indirect calorimetry in a resuscitation patient. Also, these authors raise the question of a possible use of the RQ in intensive care as an early non-invasive marker of anaerobic metabolism that can replace the invasive ones usually used (arterial lactate, venoarterial PCO2 gradient, venoarterial PCO2 gradient/ arteriovenous O2 content difference, ScVO2). However, the measurement of inspired and expired fractions in O2 and CO2 is part of the systematic monitoring of the intubated-ventilated patient in the operating room. The measurement of the VO2, VCO2 and the RQ could therefore be done from these fractions inspired and expired in O2 and CO2 by the following equation:

RQ = (FeCO2-FiCO2) / (FiO2-FeO2) The main objective of our work is to demonstrate the ability of the RQ, measured indirectly from the anesthesia ventilator, to predict the occurrence of anaerobic metabolism in patients operated of major non-cardiac surgical operation in the operating room. Secondly, the objective is to evaluate the association between the variations of the RQ, EtCO2, Dc, ScVO2, venoarterial PCO2 gradient, venoarterial PCO2 gradient/arteriovenous O2 content difference and lactate levels at different times during the surgical procedure and depending on the occurrence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the operating room of Amiens University Hospital supported for major non-cardiac surgery (abdominal, orthopedic, vascular) for which the practitioner had decided in accordance with the care protocols of the department to carry out an hemodynamic optimization,
* Patients monitored by a central venous catheter and an invasive measurement of blood pressure,
* Ventilated patients in controlled mode,
* Major patients.

Exclusion Criteria:

* Cardiac surgery with the need of extracorporeal circulation
* Thoracic surgery with the need of unipulmonary ventilation
* Permanent laparoscopic surgery and up to 30 minutes after exsufflation of CO2
* Acute or chronic respiratory insufficiency documented
* Interstitial lung disease with diffusion disorders
* Preoperative oxygen therapy
* Acute Respiratory Distress Syndrome with FiO2> 60%.
* Refusal of patient participation.
* Pregnant woman.
* Patient under guardianship or curatorship or deprived of public right.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the operating room of Amiens University Hospital supported for major non-cardiac surgery (abdominal, orthopedic, vascular) for which the practitioner had decided in accordance with the care protocols of the department to carry out an hemodynamic optimization
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Quotient (RQ) | 1 Month
  indirectly measured from the anesthetic respirator, and its predictive ability to develop anaerobic metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BAR, Dr, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens-Picardie, Amiens, France

REFERENCES:
- [Derived] Bar S, Grenez C, Nguyen M, de Broca B, Bernard E, Abou-Arab O, Bouhemad B, Lorne E, Guinot PG. Predicting postoperative complications with the respiratory exchange ratio after high-risk noncardiac surgery: A prospective cohort study. Eur J Anaesthesiol. 2020 Nov;37(11):1050-1057. doi: 10.1097/EJA.0000000000001111. PMID 31688330